CLINICAL TRIAL: NCT06770504
Title: The Safety and Efficacy of YTS109 Cell Injection for Relapsed/Refractory Autoimmune Hemolytic Anemia Patients After Receiving Three or More Lines of Therapy.
Brief Title: A Study of YTS109 Cell Injection in Subjects With Relapsed/Refractory Autoimmune Hemolytic Anemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Shi, Director of the Red Blood Cell Disorders Center & Director of the Regenerative Medicine Clinic, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YTS109-004
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Autoimmune Hemolytic Anemia; Anti-CD19 STAR T-cell Therapy; Failure ≥3 Lines of Therapies
Keywords: Relapsed/Refractory Autoimmune Hemolytic Anemia; CD19-STAR T cells
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YTS109 (Experimental): Participants will receive YTS109 cell infusion after preconditioning, and they need to be closely monitored for 24 hours following START-T cell infusion.
  Interventions: Biological: YTS109

INTERVENTIONS:
Biological: YTS109 — In this study, subjects will receive YTS109 Cell Injection(0.5-1E6 STAR+T cell/kg) once.

SUMMARY:
This is a Phase I, single-arm, open-label, dose-escalation and dose-expansion study. The primary objective is to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of YTS109 START T-cell therapy in patients with autoimmune hemolytic anemia who have failed ≥3 lines of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥12 years, regardless of gender.
* Diagnosis of AIHA or Evans syndrome [including warm antibody, mixed AIHA and cold antibody AIHA (Cold agglutinin disease)].
* Failure or intolerance to at least 3 lines of therapy: glucocorticoids and/or rituximab, and any one of the following treatments (splenectomy, cyclosporine, cyclophosphamide, azathioprine, mycophenolate mofetil, bendamustine, fludarabine, bortezomib, etc.Biologics, including anti-CD38 monoclonal antibody, BTK inhibitor, Syk inhibitor and complement inhibitor) (HGB < 100g/L).
* Adequate organ function: a. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN. b. Creatinine clearance (CrCl) (Cockcroft-Gault formula) ≥60ml/min. c.Blood oxygen saturation (SpO2) ≥92%.
* ECOG performance status≤2
* Subjects of childbearing potential will be required to follow contraception requirements from the time of enrollment until the end of the 12-month safety follow-up period.
* The subjects voluntarily participate in the study, sign the informed consent, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Diagnosis of lymphoproliferative tumor
* Other hereditary or acquired hemolytic diseases (Secondary AIHA caused by drugs or infection)
* The platelet count in peripheral blood<30×10^9/L
* Pregnant or breast-feeding subjects
* Receive any of the following treatments within the specified time before cell infusion: a.anti-CD20 monoclonal antibodies <12 weeks, b.sutimlimab or other marketed biologics <5 half-lives,c.plasma exchange <4 weeks, d.post-splenectomy <12 weeks, e. BTK inhibitors, anti-CD38 monoclonal antibody, Syk inhibitors, BAFF inhibitors < 5 half-lives.
* Previously received organ or stem cell transplantation
* History of new thrombosis or organ infarction in the past 6 months
* Diagnosis of the active stage of the connective tissue disease.
* Have active infections, such as sepsis, bacteremia, fungemia, uncontrolled pulmonary infection and active tuberculosis, etc.
* Positive hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg); positive hepatitis B e antibody (HBe-Ab) or hepatitis B core antibody (HBc-Ab), and the HBV-DNA copy number is above the lower limit of the measurable capacity; positive hepatitis C (HCV) antibody; positive human immunodeficiency virus (HIV) antibody; positive syphilis test.
* Underwent major surgery within 4 weeks before screening, as determined by the investigator to be unsuitable for enrollment.
* Have malignant tumors within 5 years before enrollment, except tumors with negligible risk of metastasis or death and curable tumors, such as adequately treated cervical carcinoma in situ, cutaneous basal cell carcinoma, etc.
* Have any of the following cardiovascular diseases: a.Left ventricular ejection fraction (LVEF) ≤45%, b. presence of active heart disease or congestive heart failure (New York Heart Association [NYHA] Class III or IV)), c.severe arrhythmias requiring treatment, d.have myocardial infarction, bypass surgery, or stent placement within the 6 months before the study, e.other heart diseases judged by the researcher to be unsuitable for enrollment.
* Have a history of live attenuated vaccines within 6 weeks before enrollment.
* Have a history of epilepsy or other active central nervous system diseases.
* Have an allergy to the ingredients of the medicine used in this study.
* Previously received CAR-T cell therapy.
* Patients considered to be ineligible for the study by the investigator for reasons other than the above.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Within 28 days after infusion
The incidence and frequency of treatment-emergent adverse events | Within 12 months after infusion
  Safety assessments are conducted using the NCI-CTCAE version 5.0 standards.
Best overall response rate (BOR) of each dose group | Within 12 weeks after infusion
  BOR is determined as the most favorable response observed after cell infusion, until either disease relapse or the completion of a specified observation period.
Objective response rate (ORR) of each dose group | Within 4 weeks after infusion
Time to response (TTR) | Within 6 months after infusion
  TTR is defined as the duration from cell infusion to the achievement of a hematological response